CLINICAL TRIAL: NCT03642782
Title: Evaluation of the Electroretinogram Pattern (Diopsys® NOVA System) for the Early Diagnosis of Glaucoma
Acronym: DIOPSYS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIOPSYS
Record Dates: First submitted 2018-08-13; First posted 2018-08-22 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
Keywords: electroretinogram pattern
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- early age of glaucoma or with important risk factors (Experimental): All patients included will benefit from a complete ophtalmic examination including visual acuity, slit lamp biomicroscopic examination of the anterior segment, measurement of intraocular pressure by Goldmann tonometer aplanation, dynamic gonioscopy with Posner glass. They will also have a fundus examination with examination of the retina, macula and optic nerve as well as the ERGP.
  Interventions: Device: Electroretinogram Pattern (Diopsys® NOVA System)

INTERVENTIONS:
Device: Electroretinogram Pattern (Diopsys® NOVA System) — it's an additional examination that extends the duration of the ophthalmological consultation by 30 minutes

SUMMARY:
Glaucoma is a common and potentially blinding disease. It is characterized by an optic nerve damage, a visual field defect and elevated intraocular pressure (IOP).

The loss of retinal nerve fibers is accompanied by functional impairment in the territories corresponding to deficits of the visual field. However, this structure-function relationship is not always found initially. These discrepancies are mainly chronological: the structural damage preceding the functional impairment sometimes of several years

DETAILED DESCRIPTION:
The electroretinogram pattern (ERGP) is an electrophysiological exploration technique that reflects the activity of retinal ganglion cells. It presents itself as an objective field of vision that does not require the active collaboration of the patient. It consists in recording the electrical activity of functional retinal ganglion cells following a light stimulation. Simple (30 minutes maximum), it could improve the detection of early forms of glaucoma. A significant ERGP is also thought to be correlated with peripapillary and macular CNP structural involvement of the ganglionic complex in early forms of glaucoma (MD> -6 dB).

Some results even suggest that ganglion dysfunction could be detected by the ERGP eight years on average before the occurrence of detectable alterations on the RNFL OCT. ERGP is already recognized as a routine examination for monitoring glaucomatous patients (review side in nomenclature and reimbursed by Social Security) but it could therefore be used as a diagnostic tool in very early forms of intraocular hypertonia glaucoma so to objectify signs of preperimetric functional impairment in order to establish a suitable hypotonizing treatment and to improve the prognosis of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Man and woman age ≥ 18 years
* Francophone
* Patient with medical insurance
* Refraction: sphere ± 5.0 D and cylinder ± 3.0 D
* Pupillary diameter ≥ 3mm
* Early glaucoma patients :

  * Intraocular pressure> 21 mmHg or <21mmHg under treatment
  * Thickness of pathological retinal nerve fibers with at least one affected area (OCT)
  * At least one reliable visual field (false positives, false negatives and fixation losses ≤ 25%) and no artifacts, with Corrected Pattern Standard Deviation (CPSD) pathological in the 5% and Glaucoma Hemifield Pathological test and an early attack (MD> -6dB)
* Patient at risk for glaucoma with:

  * And / or family history of glaucoma
  * and / or intraocular pressure> 21 mmHg
  * and / or retinal nerve fibers (pathological thickness in at least one area on the OCT)
  * and / or reliable visual field (false positives, false negatives and fixation losses ≤ 25%) and without artifact, with pathological Corrected Pattern Standard Deviation (CPSD) in the 5% and Glaucoma Hemifield Pathological Test and an early onset (MD> -6 dB).

Exclusion Criteria:

* Visual acuity below 20/30 (Snellen scale or equivalent on another visual acuity scale)
* Unreliable visual field (false positives, loss of fixation and false negatives> 25%)
* History of intraocular surgery (except uncomplicated cataract surgery)
* Ocular pathology other than associated glaucoma
* Neurological disease affecting the visual field or the optic nerve
* History of macular laser or pan retinal photocoagulation
* Unreliable ERGP pattern
* Offset OCT, unreliable
* Refusal to participate in the study
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Epileptic patient
* Eczema of the eyelids or allergy to one of the components of the electrodes or skin gel allowing the cleaning of the skin before the positioning of the electrodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlations between Electroretinogram Pattern, vision field and optical coherence tomography | Time of inclusion
  Electroretinogram Patterny : Magnitude, magnitude D, Magnitude D/Magnitude ratio.
Correlations between Electroretinogram Pattern, vision field and optical coherence | Time of inclusion
  Vision field: mean deviation, corrected pattern standard deviation.
Correlations between Electroretinogram Pattern, vision field and optical coherence | Time of inclusion
  Optical coherence tomography: retinal nerve fiber layer thickness and macular analysis of the ganglionic complex.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Gordon MO, Beiser JA, Brandt JD, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Kass MA. The Ocular Hypertension Treatment Study: baseline factors that predict the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):714-20; discussion 829-30. doi: 10.1001/archopht.120.6.714. PMID 12049575
- [Result] Quigley HA, Dunkelberger GR, Green WR. Retinal ganglion cell atrophy correlated with automated perimetry in human eyes with glaucoma. Am J Ophthalmol. 1989 May 15;107(5):453-64. doi: 10.1016/0002-9394(89)90488-1. PMID 2712129
- [Result] Harwerth RS, Quigley HA. Visual field defects and retinal ganglion cell losses in patients with glaucoma. Arch Ophthalmol. 2006 Jun;124(6):853-9. doi: 10.1001/archopht.124.6.853. PMID 16769839
- [Result] Sommer A, Katz J, Quigley HA, Miller NR, Robin AL, Richter RC, Witt KA. Clinically detectable nerve fiber atrophy precedes the onset of glaucomatous field loss. Arch Ophthalmol. 1991 Jan;109(1):77-83. doi: 10.1001/archopht.1991.01080010079037. PMID 1987954
- [Result] Hwang YH, Kim YY, Kim HK, Sohn YH. Ability of cirrus high-definition spectral-domain optical coherence tomography clock-hour, deviation, and thickness maps in detecting photographic retinal nerve fiber layer abnormalities. Ophthalmology. 2013 Jul;120(7):1380-7. doi: 10.1016/j.ophtha.2012.12.048. Epub 2013 Mar 28. PMID 23541761
- [Result] Tan O, Chopra V, Lu AT, Schuman JS, Ishikawa H, Wollstein G, Varma R, Huang D. Detection of macular ganglion cell loss in glaucoma by Fourier-domain optical coherence tomography. Ophthalmology. 2009 Dec;116(12):2305-14.e1-2. doi: 10.1016/j.ophtha.2009.05.025. Epub 2009 Sep 10. PMID 19744726
- [Result] Na JH, Lee K, Lee JR, Baek S, Yoo SJ, Kook MS. Detection of macular ganglion cell loss in preperimetric glaucoma patients with localized retinal nerve fibre defects by spectral-domain optical coherence tomography. Clin Exp Ophthalmol. 2013 Dec;41(9):870-80. doi: 10.1111/ceo.12142. Epub 2013 Jul 5. PMID 23777476
- [Result] Mwanza JC, Oakley JD, Budenz DL, Anderson DR; Cirrus Optical Coherence Tomography Normative Database Study Group. Ability of cirrus HD-OCT optic nerve head parameters to discriminate normal from glaucomatous eyes. Ophthalmology. 2011 Feb;118(2):241-8.e1. doi: 10.1016/j.ophtha.2010.06.036. Epub 2010 Oct 28. PMID 20920824
- [Result] Hwang YH, Kim YY. Glaucoma diagnostic ability of quadrant and clock-hour neuroretinal rim assessment using cirrus HD optical coherence tomography. Invest Ophthalmol Vis Sci. 2012 Apr 24;53(4):2226-34. doi: 10.1167/iovs.11-8689. PMID 22410556
- [Result] De Jong LA, Snepvangers CE, van den Berg TJ, Langerhorst CT. Blue-yellow perimetry in the detection of early glaucomatous damage. Doc Ophthalmol. 1990 Oct;75(3-4):303-14. doi: 10.1007/BF00164844. PMID 2090405
- [Result] Felius J, de Jong LA, van den Berg TJ, Greve EL. Functional characteristics of blue-on-yellow perimetric thresholds in glaucoma. Invest Ophthalmol Vis Sci. 1995 Jul;36(8):1665-74. PMID 7601646
- [Result] Sample PA, Taylor JD, Martinez GA, Lusky M, Weinreb RN. Short-wavelength color visual fields in glaucoma suspects at risk. Am J Ophthalmol. 1993 Feb 15;115(2):225-33. doi: 10.1016/s0002-9394(14)73928-5. PMID 8430733
- [Result] Anderson AJ, Johnson CA. Frequency-doubling technology perimetry. Ophthalmol Clin North Am. 2003 Jun;16(2):213-25. doi: 10.1016/s0896-1549(03)00011-7. PMID 12809159
- [Result] Anderson AJ, Johnson CA, Fingeret M, Keltner JL, Spry PG, Wall M, Werner JS. Characteristics of the normative database for the Humphrey matrix perimeter. Invest Ophthalmol Vis Sci. 2005 Apr;46(4):1540-8. doi: 10.1167/iovs.04-0968. PMID 15790927
- [Result] Artes PH, Hutchison DM, Nicolela MT, LeBlanc RP, Chauhan BC. Threshold and variability properties of matrix frequency-doubling technology and standard automated perimetry in glaucoma. Invest Ophthalmol Vis Sci. 2005 Jul;46(7):2451-7. doi: 10.1167/iovs.05-0135. PMID 15980235
- [Result] Mafei L, Fiorentini A. Electroretinographic responses to alternating gratings before and after section of the optic nerve. Science. 1981 Feb 27;211(4485):953-5. doi: 10.1126/science.7466369.
- [Result] Bowd C, Tafreshi A, Zangwill LM, Medeiros FA, Sample PA, Weinreb RN. Pattern electroretinogram association with spectral domain-OCT structural measurements in glaucoma. Eye (Lond). 2011 Feb;25(2):224-32. doi: 10.1038/eye.2010.203. Epub 2010 Dec 24. PMID 21183943
- [Result] Bowd C, Tafreshi A, Vizzeri G, Zangwill LM, Sample PA, Weinreb RN. Repeatability of pattern electroretinogram measurements using a new paradigm optimized for glaucoma detection. J Glaucoma. 2009 Aug;18(6):437-42. doi: 10.1097/IJG.0b013e31818c6f44. PMID 19680050
- [Result] Bowd C, Vizzeri G, Tafreshi A, Zangwill LM, Sample PA, Weinreb RN. Diagnostic accuracy of pattern electroretinogram optimized for glaucoma detection. Ophthalmology. 2009 Mar;116(3):437-43. doi: 10.1016/j.ophtha.2008.10.026. Epub 2009 Jan 22. PMID 19167080
- [Result] Tafreshi A, Racette L, Weinreb RN, Sample PA, Zangwill LM, Medeiros FA, Bowd C. Pattern electroretinogram and psychophysical tests of visual function for discriminating between healthy and glaucoma eyes. Am J Ophthalmol. 2010 Mar;149(3):488-95. doi: 10.1016/j.ajo.2009.09.027. PMID 20172073
- [Result] Ventura LM, Porciatti V. Restoration of retinal ganglion cell function in early glaucoma after intraocular pressure reduction: a pilot study. Ophthalmology. 2005 Jan;112(1):20-7. doi: 10.1016/j.ophtha.2004.09.002. PMID 15629815
- [Result] Bach M, Unsoeld AS, Philippin H, Staubach F, Maier P, Walter HS, Bomer TG, Funk J. Pattern ERG as an early glaucoma indicator in ocular hypertension: a long-term, prospective study. Invest Ophthalmol Vis Sci. 2006 Nov;47(11):4881-7. doi: 10.1167/iovs.05-0875. PMID 17065502
- [Result] Ventura LM, Sorokac N, De Los Santos R, Feuer WJ, Porciatti V. The relationship between retinal ganglion cell function and retinal nerve fiber thickness in early glaucoma. Invest Ophthalmol Vis Sci. 2006 Sep;47(9):3904-11. doi: 10.1167/iovs.06-0161. PMID 16936103
- [Result] Banitt MR, Ventura LM, Feuer WJ, Savatovsky E, Luna G, Shif O, Bosse B, Porciatti V. Progressive loss of retinal ganglion cell function precedes structural loss by several years in glaucoma suspects. Invest Ophthalmol Vis Sci. 2013 Mar 28;54(3):2346-52. doi: 10.1167/iovs.12-11026. PMID 23412088